CLINICAL TRIAL: NCT00004992
Title: Diabetes Prevention Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: (IND) - DPP (completed); U01DK048489 (NIH)
Record Dates: First submitted 2000-03-17; First posted 2000-03-20 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Glucose Intolerance
Keywords: clinical trial; multi-center; NIDDM; NIDDK; Diabetes Prevention Program (DPP); diabetes risk factors; diabetes; glycemia; cardiovascular risk factors; quality of life; physical activity and nutrition; occurrence of adverse events; insulin secretion and sensitivity; prevention; abnormal glucose metabolism; lifestyle intervention; drug intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Diabetes Mellitus; Motor Activity; Hypersensitivity | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Intensive Lifestyle (Active Comparator)
  Interventions: Behavioral: Intensive lifestyle

INTERVENTIONS:
Behavioral: Intensive lifestyle
  Arms: Intensive Lifestyle
Drug: Metformin
  Arms: Metformin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The Diabetes Prevention Program is a nationwide clinical study to answer the question: Can Type 2 diabetes (also called noninsulin-dependent or adult-onset diabetes) be prevented or delayed? The study has recruited volunteers, who are at high risk of developing diabetes, at twenty-five medical centers in the United States. It is sponsored by the National Institute of Diabetes and Digestive and Kidney Diseases of the National Institutes of Health, and other Institute and corporate sponsors. Researchers will evaluate the efficacy of a lifestyle intervention and a pharmacological intervention in preventing or delaying Type 2 diabetes in persons with impaired glucose tolerance (IGT). Each person in the study will be followed for 3 to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance (fasting plasma glucose 95-125 mg/dL and 2hr plasma glucose 140-199 mg/dL)
* BMI >= 24 kg/m2

Exclusion Criteria:

* Underlying disease likely to limit life span and/or increase risk of interventions
* Conditions or behaviors likely to effect conduct of the DPP
* Diabetes or disordered glucose metabolism
* Suboptimally treated Thyroid disease
* Fasting triglyceride level < 600 mg/dl
* Exclusions related to medications

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3234 (Actual)
Dates: Start 1996-07; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Development of diabetes | Up to 5 years
  Diabetes was diagnosed on the basis of an annual oral glucose-tolerance test or a semiannual fasting plasma glucose test, according to the 1997 criteria of the American Diabetes Association

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fowler, PhD, Principal Investigator — George Washington University Biostatistics Center
Locations (1):
- George Washington University Biostatistics Center, Suite 750, 6110 Executive Blvd, Rockville, Maryland, United States

REFERENCES:
- [Result] Florez JC, Jablonski KA, Bayley N, Pollin TI, de Bakker PI, Shuldiner AR, Knowler WC, Nathan DM, Altshuler D; Diabetes Prevention Program Research Group. TCF7L2 polymorphisms and progression to diabetes in the Diabetes Prevention Program. N Engl J Med. 2006 Jul 20;355(3):241-50. doi: 10.1056/NEJMoa062418. PMID 16855264
- [Result] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Derived] Lin PD, Cardenas A, Temprosa M, Botelho JC, Calafat AM, Gold DR, Oken E, Fleisch AF. Associations of Perfluoroalkyl and Polyfluoroalkyl Substances With Cardiovascular Disease Incidence in Adults With Prediabetes: Findings From the Diabetes Prevention Program. J Am Heart Assoc. 2026 Jan 6;15(1):e046298. doi: 10.1161/JAHA.125.046298. Epub 2025 Dec 18. PMID 41413398
- [Derived] Tjaden AH, Goldbaum AA, Edelstein SL, Heckman-Stoddard BM, Reedy J, Herman WH, Hoskin M, Knowler WC, Schlogl M, Temple KA, Venditti EM, Watson K, Temprosa M, Shams-White MM; DPP Research Group. The 2018 World Cancer Research Fund/American Institute for Cancer Research Score and Cancer Risk: results from the diabetes prevention program outcomes study. Am J Clin Nutr. 2025 Sep;122(3):715-723. doi: 10.1016/j.ajcnut.2025.07.011. Epub 2025 Jul 15. PMID 40675492
- [Derived] Knowler WC, Doherty L, Edelstein SL, Bennett PH, Dabelea D, Hoskin M, Kahn SE, Kalyani RR, Kim C, Pi-Sunyer FX, Raghavan S, Shah VO, Temprosa M, Venditti EM, Nathan DM; DPP/DPPOS Research Group. Long-term effects and effect heterogeneity of lifestyle and metformin interventions on type 2 diabetes incidence over 21 years in the US Diabetes Prevention Program randomised clinical trial. Lancet Diabetes Endocrinol. 2025 Jun;13(6):469-481. doi: 10.1016/S2213-8587(25)00022-1. Epub 2025 Apr 28. PMID 40311647
- [Derived] Munshi MN, Venditti EM, Tjaden AH, Knowler WC, Boyko EJ, Middelbeek RJW, Luchsinger JA, Lee CG, Hazuda HP, Salive ME, Edelstein SL, Storer TW. Long-term impact of Diabetes Prevention Program interventions on walking endurance. Front Public Health. 2024 Dec 18;12:1470035. doi: 10.3389/fpubh.2024.1470035. eCollection 2024. PMID 39744353
- [Derived] Molitch ME, Tripputi M, Levey AS, Crandall JP, Dabelea D, Herman WH, Knowler WC, Orchard TJ, Schroeder EB, Srikanthan P, Temprosa M, White NH, Nathan DM; Diabetes Prevention Program Research Group. Electronic address: dppmail@bsc.gwu.edu. Effects of metformin and intensive lifestyle interventions on the incidence of kidney disease in adults in the DPP/DPPOS. J Diabetes Complications. 2023 Sep;37(9):108556. doi: 10.1016/j.jdiacomp.2023.108556. Epub 2023 Jul 25. PMID 37607422
- [Derived] Shams-White MM, Tjaden AH, Edelstein SL, Bassiouni S, Kahle LL, Kim C, Pi-Sunyer X, Temple KA, Venditti EM, Reedy J, Heckman-Stoddard BM; DPP Research Group. The 2018 World Cancer Research Fund (WCRF)/American Institute for Cancer Research (AICR) score and diabetes risk in the Diabetes Prevention Program Outcomes Study (DPPOS). BMC Nutr. 2022 Sep 21;8(1):105. doi: 10.1186/s40795-022-00596-7. PMID 36131333
- [Derived] Vazquez Arreola E, Knowler WC, Hanson RL. Weight Loss, Lifestyle Intervention, and Metformin Affect Longitudinal Relationship of Insulin Secretion and Sensitivity. J Clin Endocrinol Metab. 2022 Nov 23;107(11):3086-3099. doi: 10.1210/clinem/dgac509. PMID 36062951
- [Derived] Goldberg RB, Orchard TJ, Crandall JP, Boyko EJ, Budoff M, Dabelea D, Gadde KM, Knowler WC, Lee CG, Nathan DM, Watson K, Temprosa M; Diabetes Prevention Program Research Group*. Effects of Long-term Metformin and Lifestyle Interventions on Cardiovascular Events in the Diabetes Prevention Program and Its Outcome Study. Circulation. 2022 May 31;145(22):1632-1641. doi: 10.1161/CIRCULATIONAHA.121.056756. Epub 2022 May 23. PMID 35603600
- [Derived] Wander PL, Christophi CA, Araneta MRG, Boyko EJ, Enquobahrie DA, Dabelea D, Goldberg RB, Kahn SE, Kim C, Pi-Sunyer X, Knowler WC. Adiposity, related biomarkers, and type 2 diabetes after gestational diabetes: The Diabetes Prevention Program. Obesity (Silver Spring). 2022 Jan;30(1):221-228. doi: 10.1002/oby.23291. Epub 2021 Nov 18. PMID 34796678
- [Derived] Lee CG, Heckman-Stoddard B, Dabelea D, Gadde KM, Ehrmann D, Ford L, Prorok P, Boyko EJ, Pi-Sunyer X, Wallia A, Knowler WC, Crandall JP, Temprosa M; Diabetes Prevention Program Research Group; Diabetes Prevention Program Research Group:. Effect of Metformin and Lifestyle Interventions on Mortality in the Diabetes Prevention Program and Diabetes Prevention Program Outcomes Study. Diabetes Care. 2021 Dec;44(12):2775-2782. doi: 10.2337/dc21-1046. Epub 2021 Oct 25. PMID 34697033
- [Derived] Varga TV, Liu J, Goldberg RB, Chen G, Dagogo-Jack S, Lorenzo C, Mather KJ, Pi-Sunyer X, Brunak S, Temprosa M; Diabetes Prevention Program Research Group. Predictive utilities of lipid traits, lipoprotein subfractions and other risk factors for incident diabetes: a machine learning approach in the Diabetes Prevention Program. BMJ Open Diabetes Res Care. 2021 Mar;9(1):e001953. doi: 10.1136/bmjdrc-2020-001953. PMID 33789908
- [Derived] Goldberg RB, Tripputi MT, Boyko EJ, Budoff M, Chen ZZ, Clark JM, Dabelea DM, Edelstein SL, Gerszten RE, Horton E, Mather KJ, Perreault L, Temprosa M, Wallia A, Watson K, Irfan Z. Hepatic Fat in Participants With and Without Incident Diabetes in the Diabetes Prevention Program Outcome Study. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4746-e4765. doi: 10.1210/clinem/dgab160. PMID 33705543
- [Derived] Kriska AM, Rockette-Wagner B, Edelstein SL, Bray GA, Delahanty LM, Hoskin MA, Horton ES, Venditti EM, Knowler WC; DPP Research Group. The Impact of Physical Activity on the Prevention of Type 2 Diabetes: Evidence and Lessons Learned From the Diabetes Prevention Program, a Long-Standing Clinical Trial Incorporating Subjective and Objective Activity Measures. Diabetes Care. 2021 Jan;44(1):43-49. doi: 10.2337/dc20-1129. Epub 2020 Nov 10. PMID 33444158
- [Derived] Hazuda HP, Pan Q, Florez H, Luchsinger JA, Crandall JP, Venditti EM, Golden SH, Kriska AM, Bray GA. Association of Intensive Lifestyle and Metformin Interventions With Frailty in the Diabetes Prevention Program Outcomes Study. J Gerontol A Biol Sci Med Sci. 2021 Apr 30;76(5):929-936. doi: 10.1093/gerona/glaa295. PMID 33428709
- [Derived] Gupta DK, Walford GA, Ma Y, Jarolim P, Wang TJ; DPP Research Group. Racial/ethnic differences in circulating natriuretic peptide levels: The Diabetes Prevention Program. PLoS One. 2020 Feb 21;15(2):e0229280. doi: 10.1371/journal.pone.0229280. eCollection 2020. PMID 32084251
- [Derived] Merino J, Jablonski KA, Mercader JM, Kahn SE, Chen L, Harden M, Delahanty LM, Araneta MRG, Walford GA, Jacobs SBR, Ibebuogu UN, Franks PW, Knowler WC, Florez JC; Diabetes Prevention Program Research Group. Interaction Between Type 2 Diabetes Prevention Strategies and Genetic Determinants of Coronary Artery Disease on Cardiometabolic Risk Factors. Diabetes. 2020 Jan;69(1):112-120. doi: 10.2337/db19-0097. Epub 2019 Oct 21. PMID 31636172
- [Derived] Perreault L, Pan Q, Schroeder EB, Kalyani RR, Bray GA, Dagogo-Jack S, White NH, Goldberg RB, Kahn SE, Knowler WC, Mathioudakis N, Dabelea D; Diabetes Prevention Program Research Group. Regression From Prediabetes to Normal Glucose Regulation and Prevalence of Microvascular Disease in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabetes Care. 2019 Sep;42(9):1809-1815. doi: 10.2337/dc19-0244. Epub 2019 Jul 18. PMID 31320445
- [Derived] Cardenas A, Hivert MF, Gold DR, Hauser R, Kleinman KP, Lin PD, Fleisch AF, Calafat AM, Ye X, Webster TF, Horton ES, Oken E. Associations of Perfluoroalkyl and Polyfluoroalkyl Substances With Incident Diabetes and Microvascular Disease. Diabetes Care. 2019 Sep;42(9):1824-1832. doi: 10.2337/dc18-2254. Epub 2019 Jul 11. PMID 31296647
- [Derived] Apolzan JW, Venditti EM, Edelstein SL, Knowler WC, Dabelea D, Boyko EJ, Pi-Sunyer X, Kalyani RR, Franks PW, Srikanthan P, Gadde KM; Diabetes Prevention Program Research Group. Long-Term Weight Loss With Metformin or Lifestyle Intervention in the Diabetes Prevention Program Outcomes Study. Ann Intern Med. 2019 May 21;170(10):682-690. doi: 10.7326/M18-1605. Epub 2019 Apr 23. PMID 31009939
- [Derived] Diabetes Prevention Program Research Group. Long-term Effects of Metformin on Diabetes Prevention: Identification of Subgroups That Benefited Most in the Diabetes Prevention Program and Diabetes Prevention Program Outcomes Study. Diabetes Care. 2019 Apr;42(4):601-608. doi: 10.2337/dc18-1970. PMID 30877090
- [Derived] Cardenas A, Hauser R, Gold DR, Kleinman KP, Hivert MF, Fleisch AF, Lin PD, Calafat AM, Webster TF, Horton ES, Oken E. Association of Perfluoroalkyl and Polyfluoroalkyl Substances With Adiposity. JAMA Netw Open. 2018 Aug 3;1(4):e181493. doi: 10.1001/jamanetworkopen.2018.1493. PMID 30646133
- [Derived] Hivert MF, Christophi CA, Jablonski KA, Edelstein SL, Kahn SE, Golden SH, Dagogo-Jack S, Mather KJ, Luchsinger JA, Caballero AE, Barrett-Connor E, Knowler WC, Florez JC, Herman WH. Genetic Ancestry Markers and Difference in A1c Between African American and White in the Diabetes Prevention Program. J Clin Endocrinol Metab. 2019 Feb 1;104(2):328-336. doi: 10.1210/jc.2018-01416. PMID 30358859
- [Derived] DeBoer MD, Filipp SL, Gurka MJ. Use of a Metabolic Syndrome Severity Z Score to Track Risk During Treatment of Prediabetes: An Analysis of the Diabetes Prevention Program. Diabetes Care. 2018 Nov;41(11):2421-2430. doi: 10.2337/dc18-1079. Epub 2018 Oct 1. PMID 30275282
- [Derived] Berger SE, Huggins GS, McCaffery JM, Lichtenstein AH. Comparison among criteria to define successful weight-loss maintainers and regainers in the Action for Health in Diabetes (Look AHEAD) and Diabetes Prevention Program trials. Am J Clin Nutr. 2017 Dec;106(6):1337-1346. doi: 10.3945/ajcn.117.157446. Epub 2017 Oct 18. PMID 29046304
- [Derived] Herman WH, Pan Q, Edelstein SL, Mather KJ, Perreault L, Barrett-Connor E, Dabelea DM, Horton E, Kahn SE, Knowler WC, Lorenzo C, Pi-Sunyer X, Venditti E, Ye W; Diabetes Prevention Program Research Group. Impact of Lifestyle and Metformin Interventions on the Risk of Progression to Diabetes and Regression to Normal Glucose Regulation in Overweight or Obese People With Impaired Glucose Regulation. Diabetes Care. 2017 Dec;40(12):1668-1677. doi: 10.2337/dc17-1116. Epub 2017 Oct 11. PMID 29021207
- [Derived] Sylvetsky AC, Edelstein SL, Walford G, Boyko EJ, Horton ES, Ibebuogu UN, Knowler WC, Montez MG, Temprosa M, Hoskin M, Rother KI, Delahanty LM; Diabetes Prevention Program Research Group. A High-Carbohydrate, High-Fiber, Low-Fat Diet Results in Weight Loss among Adults at High Risk of Type 2 Diabetes. J Nutr. 2017 Nov;147(11):2060-2066. doi: 10.3945/jn.117.252395. Epub 2017 Sep 27. PMID 28954840
- [Derived] Perreault L, Pan Q, Aroda VR, Barrett-Connor E, Dabelea D, Dagogo-Jack S, Hamman RF, Kahn SE, Mather KJ, Knowler WC; Diabetes Prevention Program Research Group. Exploring residual risk for diabetes and microvascular disease in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabet Med. 2017 Dec;34(12):1747-1755. doi: 10.1111/dme.13453. Epub 2017 Sep 19. PMID 28833481
- [Derived] Aroda VR, Knowler WC, Crandall JP, Perreault L, Edelstein SL, Jeffries SL, Molitch ME, Pi-Sunyer X, Darwin C, Heckman-Stoddard BM, Temprosa M, Kahn SE, Nathan DM; Diabetes Prevention Program Research Group. Metformin for diabetes prevention: insights gained from the Diabetes Prevention Program/Diabetes Prevention Program Outcomes Study. Diabetologia. 2017 Sep;60(9):1601-1611. doi: 10.1007/s00125-017-4361-9. Epub 2017 Aug 2. PMID 28770322
- [Derived] Herman WH. The cost-effectiveness of diabetes prevention: results from the Diabetes Prevention Program and the Diabetes Prevention Program Outcomes Study. Clin Diabetes Endocrinol. 2015 Sep 2;1:9. doi: 10.1186/s40842-015-0009-1. eCollection 2015. PMID 28702228
- [Derived] Luchsinger JA, Ma Y, Christophi CA, Florez H, Golden SH, Hazuda H, Crandall J, Venditti E, Watson K, Jeffries S, Manly JJ, Pi-Sunyer FX; Diabetes Prevention Program Research Group. Metformin, Lifestyle Intervention, and Cognition in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2017 Jul;40(7):958-965. doi: 10.2337/dc16-2376. Epub 2017 May 12. PMID 28500216
- [Derived] Varga TV, Winters AH, Jablonski KA, Horton ES, Khare-Ranade P, Knowler WC, Marcovina SM, Renstrom F, Watson KE, Goldberg R, Florez JC, Pollin TI, Franks PW. Comprehensive Analysis of Established Dyslipidemia-Associated Loci in the Diabetes Prevention Program. Circ Cardiovasc Genet. 2016 Dec;9(6):495-503. doi: 10.1161/CIRCGENETICS.116.001457. Epub 2016 Oct 26. PMID 27784733
- [Derived] McCaffery JM, Jablonski KA, Franks PW, Delahanty LM, Aroda V, Marrero D, Hamman RF, Horton ES, Dagogo-Jack S, Wylie-Rosett J, Barrett-Connor E, Kitabchi A, Knowler WC, Wing RR, Florez JC; Diabetes Prevention Program Research Group. Replication of the Association of BDNF and MC4R Variants With Dietary Intake in the Diabetes Prevention Program. Psychosom Med. 2017 Feb/Mar;79(2):224-233. doi: 10.1097/PSY.0000000000000380. PMID 27551991
- [Derived] Kim C, Barrett-Connor E, Aroda VR, Mather KJ, Christophi CA, Horton ES, Pi-Sunyer X, Bray GA, Labrie F, Golden SH; Diabetes Prevention Program Research Group. Testosterone and depressive symptoms among men in the Diabetes Prevention Program. Psychoneuroendocrinology. 2016 Oct;72:63-71. doi: 10.1016/j.psyneuen.2016.06.009. Epub 2016 Jun 15. PMID 27371769
- [Derived] Walford GA, Ma Y, Clish C, Florez JC, Wang TJ, Gerszten RE; Diabetes Prevention Program Research Group. Metabolite Profiles of Diabetes Incidence and Intervention Response in the Diabetes Prevention Program. Diabetes. 2016 May;65(5):1424-33. doi: 10.2337/db15-1063. Epub 2016 Feb 9. PMID 26861782
- [Derived] Papandonatos GD, Pan Q, Pajewski NM, Delahanty LM, Peter I, Erar B, Ahmad S, Harden M, Chen L, Fontanillas P; GIANT Consortium; Wagenknecht LE, Kahn SE, Wing RR, Jablonski KA, Huggins GS, Knowler WC, Florez JC, McCaffery JM, Franks PW; Diabetes Prevention Program and the Look AHEAD Research Groups. Genetic Predisposition to Weight Loss and Regain With Lifestyle Intervention: Analyses From the Diabetes Prevention Program and the Look AHEAD Randomized Controlled Trials. Diabetes. 2015 Dec;64(12):4312-21. doi: 10.2337/db15-0441. Epub 2015 Aug 7. PMID 26253612
- [Derived] Mather KJ, Kim C, Christophi CA, Aroda VR, Knowler WC, Edelstein SE, Florez JC, Labrie F, Kahn SE, Goldberg RB, Barrett-Connor E; Diabetes Prevention Program. Steroid Sex Hormones, Sex Hormone-Binding Globulin, and Diabetes Incidence in the Diabetes Prevention Program. J Clin Endocrinol Metab. 2015 Oct;100(10):3778-86. doi: 10.1210/jc.2015-2328. Epub 2015 Jul 22. PMID 26200237
- [Derived] Rockette-Wagner B, Edelstein S, Venditti EM, Reddy D, Bray GA, Carrion-Petersen ML, Dabelea D, Delahanty LM, Florez H, Franks PW, Montez MG, Rubin R, Kriska AM; Diabetes Prevention Program Research Group. The impact of lifestyle intervention on sedentary time in individuals at high risk of diabetes. Diabetologia. 2015 Jun;58(6):1198-202. doi: 10.1007/s00125-015-3565-0. Epub 2015 Apr 8. PMID 25851102
- [Derived] Marrero DG, Ma Y, de Groot M, Horton ES, Price DW, Barrett-Connor E, Carnethon MR, Knowler WC; Diabetes Prevention Program Research Group. Depressive symptoms, antidepressant medication use, and new onset of diabetes in participants of the diabetes prevention program and the diabetes prevention program outcomes study. Psychosom Med. 2015 Apr;77(3):303-10. doi: 10.1097/PSY.0000000000000156. PMID 25775165
- [Derived] Aroda VR, Christophi CA, Edelstein SL, Zhang P, Herman WH, Barrett-Connor E, Delahanty LM, Montez MG, Ackermann RT, Zhuo X, Knowler WC, Ratner RE; Diabetes Prevention Program Research Group. The effect of lifestyle intervention and metformin on preventing or delaying diabetes among women with and without gestational diabetes: the Diabetes Prevention Program outcomes study 10-year follow-up. J Clin Endocrinol Metab. 2015 Apr;100(4):1646-53. doi: 10.1210/jc.2014-3761. Epub 2015 Feb 23. PMID 25706240
- [Derived] Diabetes Prevention Program Research Group. HbA1c as a predictor of diabetes and as an outcome in the diabetes prevention program: a randomized clinical trial. Diabetes Care. 2015 Jan;38(1):51-8. doi: 10.2337/dc14-0886. Epub 2014 Oct 21. PMID 25336746
- [Derived] Diabetes Prevention Program (DPP) Research Group; Hamman RF, Horton E, Barrett-Connor E, Bray GA, Christophi CA, Crandall J, Florez JC, Fowler S, Goldberg R, Kahn SE, Knowler WC, Lachin JM, Murphy MB, Venditti E. Factors affecting the decline in incidence of diabetes in the Diabetes Prevention Program Outcomes Study (DPPOS). Diabetes. 2015 Mar;64(3):989-98. doi: 10.2337/db14-0333. Epub 2014 Oct 2. PMID 25277389
- [Derived] Franks PW, Christophi CA, Jablonski KA, Billings LK, Delahanty LM, Horton ES, Knowler WC, Florez JC; Diabetes Prevention Program Research Group. Common variation at PPARGC1A/B and change in body composition and metabolic traits following preventive interventions: the Diabetes Prevention Program. Diabetologia. 2014 Mar;57(3):485-90. doi: 10.1007/s00125-013-3133-4. Epub 2013 Dec 7. PMID 24317794
- [Derived] Goldberg R, Temprosa M, Otvos J, Brunzell J, Marcovina S, Mather K, Arakaki R, Watson K, Horton E, Barrett-Connor E. Lifestyle and metformin treatment favorably influence lipoprotein subfraction distribution in the Diabetes Prevention Program. J Clin Endocrinol Metab. 2013 Oct;98(10):3989-98. doi: 10.1210/jc.2013-1452. Epub 2013 Aug 26. PMID 23979954
- [Derived] Maruthur NM, Ma Y, Delahanty LM, Nelson JA, Aroda V, White NH, Marrero D, Brancati FL, Clark JM; Diabetes Prevention Program Research Group. Early response to preventive strategies in the Diabetes Prevention Program. J Gen Intern Med. 2013 Dec;28(12):1629-36. doi: 10.1007/s11606-013-2548-4. Epub 2013 Jul 17. PMID 23860722
- [Derived] Marrero D, Pan Q, Barrett-Connor E, de Groot M, Zhang P, Percy C, Florez H, Ackermann R, Montez M, Rubin RR; DPPOS Research Group. Impact of diagnosis of diabetes on health-related quality of life among high risk individuals: the Diabetes Prevention Program outcomes study. Qual Life Res. 2014 Feb;23(1):75-88. doi: 10.1007/s11136-013-0436-3. Epub 2013 May 26. PMID 23709097
- [Derived] Delahanty LM, Peyrot M, Shrader PJ, Williamson DA, Meigs JB, Nathan DM; DPP Research Group. Pretreatment, psychological, and behavioral predictors of weight outcomes among lifestyle intervention participants in the Diabetes Prevention Program (DPP). Diabetes Care. 2013 Jan;36(1):34-40. doi: 10.2337/dc12-0733. Epub 2012 Nov 5. PMID 23129133
- [Derived] Price DW, Ma Y, Rubin RR, Perreault L, Bray GA, Marrero D, Knowler WC, Barrett-Connor E, Lacoursiere DY; Diabetes Prevention Program Research Group. Depression as a predictor of weight regain among successful weight losers in the diabetes prevention program. Diabetes Care. 2013 Feb;36(2):216-21. doi: 10.2337/dc12-0293. Epub 2012 Sep 21. PMID 23002085
- [Derived] Florez JC, Jablonski KA, Taylor A, Mather K, Horton E, White NH, Barrett-Connor E, Knowler WC, Shuldiner AR, Pollin TI; Diabetes Prevention Program Research Group. The C allele of ATM rs11212617 does not associate with metformin response in the Diabetes Prevention Program. Diabetes Care. 2012 Sep;35(9):1864-7. doi: 10.2337/dc11-2301. Epub 2012 Jun 29. PMID 22751958
- [Derived] Florez H, Pan Q, Ackermann RT, Marrero DG, Barrett-Connor E, Delahanty L, Kriska A, Saudek CD, Goldberg RB, Rubin RR; Diabetes Prevention Program Research Group. Impact of lifestyle intervention and metformin on health-related quality of life: the diabetes prevention program randomized trial. J Gen Intern Med. 2012 Dec;27(12):1594-601. doi: 10.1007/s11606-012-2122-5. Epub 2012 Jun 13. PMID 22692637
- [Derived] Perreault L, Pan Q, Mather KJ, Watson KE, Hamman RF, Kahn SE; Diabetes Prevention Program Research Group. Effect of regression from prediabetes to normal glucose regulation on long-term reduction in diabetes risk: results from the Diabetes Prevention Program Outcomes Study. Lancet. 2012 Jun 16;379(9833):2243-51. doi: 10.1016/S0140-6736(12)60525-X. Epub 2012 Jun 9. PMID 22683134
- [Derived] Mather KJ, Christophi CA, Jablonski KA, Knowler WC, Goldberg RB, Kahn SE, Spector T, Dastani Z, Waterworth D, Richards JB, Funahashi T, Pi-Sunyer FX, Pollin TI, Florez JC, Franks PW; Diabetes Prevention Program Research Group. Common variants in genes encoding adiponectin (ADIPOQ) and its receptors (ADIPOR1/2), adiponectin concentrations, and diabetes incidence in the Diabetes Prevention Program. Diabet Med. 2012 Dec;29(12):1579-88. doi: 10.1111/j.1464-5491.2012.03662.x. PMID 22443353
- [Derived] Diabetes Prevention Program Research Group. Long-term safety, tolerability, and weight loss associated with metformin in the Diabetes Prevention Program Outcomes Study. Diabetes Care. 2012 Apr;35(4):731-7. doi: 10.2337/dc11-1299. PMID 22442396
- [Derived] Diabetes Prevention Program Research Group. The 10-year cost-effectiveness of lifestyle intervention or metformin for diabetes prevention: an intent-to-treat analysis of the DPP/DPPOS. Diabetes Care. 2012 Apr;35(4):723-30. doi: 10.2337/dc11-1468. PMID 22442395
- [Derived] Delahanty LM, Pan Q, Jablonski KA, Watson KE, McCaffery JM, Shuldiner A, Kahn SE, Knowler WC, Florez JC, Franks PW; Diabetes Prevention Program Research Group. Genetic predictors of weight loss and weight regain after intensive lifestyle modification, metformin treatment, or standard care in the Diabetes Prevention Program. Diabetes Care. 2012 Feb;35(2):363-6. doi: 10.2337/dc11-1328. Epub 2011 Dec 16. PMID 22179955
- [Derived] Florez H, Ma Y, Crandall JP, Perreault L, Marcovina SM, Bray GA, Saudek CD, Barrett-Connor E, Knowler WC; Diabetes Prevention Program Research Group. Parental longevity and diabetes risk in the Diabetes Prevention Program. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1211-7. doi: 10.1093/gerona/glr114. Epub 2011 Aug 17. PMID 21852284
- [Derived] Jablonski KA, McAteer JB, de Bakker PI, Franks PW, Pollin TI, Hanson RL, Saxena R, Fowler S, Shuldiner AR, Knowler WC, Altshuler D, Florez JC; Diabetes Prevention Program Research Group. Common variants in 40 genes assessed for diabetes incidence and response to metformin and lifestyle intervention in the diabetes prevention program. Diabetes. 2010 Oct;59(10):2672-81. doi: 10.2337/db10-0543. Epub 2010 Aug 3. PMID 20682687
- [Derived] Goldberg RB, Temprosa M, Haffner S, Orchard TJ, Ratner RE, Fowler SE, Mather K, Marcovina S, Saudek C, Matulik MJ, Price D; Diabetes Prevention Program Research Group. Effect of progression from impaired glucose tolerance to diabetes on cardiovascular risk factors and its amelioration by lifestyle and metformin intervention: the Diabetes Prevention Program randomized trial by the Diabetes Prevention Program Research Group. Diabetes Care. 2009 Apr;32(4):726-32. doi: 10.2337/dc08-0494. Epub 2009 Jan 26. PMID 19171717
- [Derived] Diabetes Prevention Program Research Group. Changes in albumin excretion in the diabetes prevention program. Diabetes Care. 2009 Apr;32(4):720-5. doi: 10.2337/dc08-1400. Epub 2009 Jan 8. PMID 19131464
- [Derived] Franks PW, Jablonski KA, Delahanty LM, McAteer JB, Kahn SE, Knowler WC, Florez JC; Diabetes Prevention Program Research Group. Assessing gene-treatment interactions at the FTO and INSIG2 loci on obesity-related traits in the Diabetes Prevention Program. Diabetologia. 2008 Dec;51(12):2214-23. doi: 10.1007/s00125-008-1158-x. Epub 2008 Oct 7. PMID 18839134
- [Derived] Moore AF, Jablonski KA, McAteer JB, Saxena R, Pollin TI, Franks PW, Hanson RL, Shuldiner AR, Knowler WC, Altshuler D, Florez JC; Diabetes Prevention Program Research Group. Extension of type 2 diabetes genome-wide association scan results in the diabetes prevention program. Diabetes. 2008 Sep;57(9):2503-10. doi: 10.2337/db08-0284. Epub 2008 Jun 10. PMID 18544707
- [Derived] Franks PW, Jablonski KA, Delahanty L, Hanson RL, Kahn SE, Altshuler D, Knowler WC, Florez JC; Diabetes Prevention Program Research Group. The Pro12Ala variant at the peroxisome proliferator-activated receptor gamma gene and change in obesity-related traits in the Diabetes Prevention Program. Diabetologia. 2007 Dec;50(12):2451-60. doi: 10.1007/s00125-007-0826-6. Epub 2007 Sep 27. PMID 17898990